CLINICAL TRIAL: NCT01789112
Title: Acute Neurotrophic Effects of a Non Excitatory Cardial Stimulation by Optimizer III System in Patients With Heart Failure
Brief Title: Acute Effects of a Non Excitatory Cardial Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-032
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: CCM Implantation
MeSH Terms: interventions — Blood Specimen Collection

ARMS (1):
- CCM aggregate (Experimental): Taking of 10 blood samples
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Taking of blood sample

SUMMARY:
Electric stimulation by cardial contractility modulation (CCM)to improve contractility and physical capacity

ELIGIBILITY:
Inclusion Criteria:

* planned CCM Implantation
* systolic left ventricular dysfunction despite of adequate therapy of heart failure (NYHA II, III, IV)
* implanted pacemaker, defibrillator or pacemaker during CS intubation
* written informed consent
* open entryways

Exclusion Criteria:

* anemia Hemoglobin (HB)<8 mg/dl
* lying coronary sinus (CS) tube or CS being not able to intubate
* chronic atrial fibrillation or flutter
* mechanic tricuspid valve prothesis
* no access via subclavian vein
* patients with VVI pacemaker being stimulated 110%
* idiopathic hypertrophic cardiomyopathy, restrictive constrictive cardiomyopathy or heart failure because of known inflammatory or infiltrative illnesses or constrictive illness
* acute myocardial ischemia presented by angina pectoris or ECG changes under load
* patients being hospitalized because of heart failure during the last month and have to be treated with intravenous diuretics or inotropic substances
* acute coronary syndrome should not be implanted for at least 3 month
* patients with mechanic aortic or tricuspid valve
* patients after heart transplantation
* patients with clinical significant ectopy, defined by > 8.900 PVCs during 24 hours at beginning Holter monitoring
* patients after hypertensive crisis
* patients with acute renal failure
* Ejection Fraction (EF) > 35
* patients after left ventricular pacemaker electrode
* pregnant or breast feeding women
* patients with heart failure after sepsis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
positive inotropic effects by CCM stimulation | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Reith, MD, Principal Investigator — RWTH Aachen, Medical Departement I Univerity Hospital Aachen
Locations (1):
- Univeristy Hospital Aachen, Aachen, North Rhine Westfalia, Germany